CLINICAL TRIAL: NCT07163000
Title: Earlier Diagnosis of Peripheral Neuropathy Using A Simple sCreening Tool (ACT)
Acronym: ACT
Status: Active, not recruiting | Type: Observational
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Procter and Gamble (Industry); Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-00029
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Neuropathy; Painful Neuropathy; Diabetes (DM)
Keywords: Diabetes; Peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuropathy, Painful; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is looking at people with diabetes (type 1 and type 2 diabetes) to see how well a short questionnaire, called the ACT, can identify nerve damage in the feet and legs (also known as peripheral neuropathy). The investigators will compare the ACT questionnaire to other commonly used tools (the DN4 and Michigan Neuropathy Screening Instrument) and to an eye-test that detects small nerve fibers in the eye (called corneal confocal microscopy, or CCM).

The main goal is to find out if the ACT questionnaire is accurate in detecting nerve damage and painful nerve damage caused by diabetes.

The investigators will also look at whether changes in blood sugar levels, measured with a continuous glucose monitor (Freestyle Libre 3 and iCan), are linked to nerve pain and small nerve fiber damage.

DETAILED DESCRIPTION:
This a cross-sectional cohort study in patients with diabetes with the aim of assessing the validity and diagnostic accuracy of the ACT questionnaire in identifying peripheral neuropathy (PN) in patients with diabetes and explore underlying mechanisms for nerve damage. The primary endpoint is to validate the ACT tool in identifying diabetic painful neuropathy against the DN4 questionnaire, Michigan Neuropathy Screening Instrument (MNSI) and in relation to underlying small nerve fibre damage (CCM). And the secondary endpoints include the investigation of the association between glycemic indices using continuous glucose monitoring (CGM- Freestyle Libre 3 and iCan) with neuropathic pain (ACT/DN4/MNSI) and small nerve fibre damage (CCM).

Participants will attend 3 visits and the following will be assessed:

* Visit 1(baseline): Consent, screening, CCM, ACT, MNSI, DN4, CGM (Freestyle Libre 3).
* Visit 2 (14-days follow-up): CGM (freestyle Libre 3), ACT, MNSI, DN4
* Visit 3 (between 1-6 months): CGM (iCan)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes (T1DM and T2DM)
* Age ≥18
* Able to provide consent.
* Able to sit still for corneal confocal microscopy

Exclusion Criteria:

* Failure to provide informed consent
* Participants with a history of ocular trauma or previous ocular surgery in the preceding 6 months, are allergic to oxybuprocaine or local anesthetics or unable to cooperate by holding still or placing their chin on an optical device
* Other causes of peripheral neuropathy: vitamin B12 deficiency; hypothyroidism; myeloma.
* Cognitively impaired participants
* Pregnant women
* Nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants attending the outpatients clinic at the diabetes center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-05-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Validation of the ACT tool | Baseline (Day 1) and then 14 days after visit 1
  Identification of number of participants with diabetic peripheral neuropathy as assessed by the ACT tool.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Rayaz A. Malik, PhD, Principal Investigator — Weill Cornell Medicine - Qatar
Locations (1):
- Weill Cornell Medicine-Qatar, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
The findings of this study will be disseminated both locally, within Qatar, and internationally through presentations at scientific conferences and publications in peer-reviewed journals. De-identified study data may be made available to qualified researchers and clinicians with a legitimate academic interest in peripheral neuropathy. Any data shared externally will be fully coded to exclude protected health information and will be subject to appropriate data-sharing agreements, such as a data use agreement, in accordance with applicable regulations and institutional policies.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the de-identified data will be accessible for 1 year, with possible extensions considered.
Access Criteria: Access to the research data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of data sharing agreement.